CLINICAL TRIAL: NCT06710067
Title: Observational Study of Urine Metabolites in the Diagnosis of Disease
Brief Title: Urine Metabolites in the Diagnosis of Disease
Status: Recruiting | Type: Observational
Sponsor: Luventix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Luventix-001; 20242000 (Other: WCG IRB)
Record Dates: First submitted 2024-09-27; First posted 2024-11-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Small Intestinal Bacterial Overgrowth Syndrome (SIBO); Crohn Disease; Celiac Disease
MeSH Terms: conditions — Colorectal Neoplasms; Crohn Disease; Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Disease Cohort

SUMMARY:
The goal of this observational study is to validate a non-invasive, urine-based diagnostic technology for the detection and differentiation of various gastrointestinal (GI) diseases.

This research study intends to enroll participants across a range of demographics and GI disease states including colorectal cancer, small intestinal bacterial overgrowth (SIBO), Crohn's disease, and Celiac disease, collect urine samples and clinical data, and use artificial intelligence and machine learning to build disease-specific models which can identify and differentiate a participants' specific GI disease.

The main questions it aims to answer are:

1. Does the platform identify a disease signal within each disease cohort, compared to normal controls?
2. How well does the test perform (e.g. sensitivity and specificity/false-positive rate)?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at time of enrollment.
* Able and willing to provide a one-time urine sample and comply with all study procedures for the study.
* Able to understand the study procedures, able to provide consent to participate in the study, and willing to authorize release of relevant protected health information by consenting to a HIPAA medical release form.

Exclusion Criteria:

* Known to be pregnant.
* A medical condition which, in the opinion of the Investigator and/or Sponsor, should preclude enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited in the United States and/or internationally, with the following order of priority and preference: ·
  1. multi-center recruitment and eligibility screen at approximately 5-10 clinical sites, and/or
  2. clinical research organization (CRO) recruitment and eligibility screen, which may include internationally recruited patients and/or
  3. decentralized recruitment via social media sites directing to an online eligibility screen and/or
  4. Biobank/biorepository sourced frozen samples
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Disease signal detection | From date of enrollment to the end of sample analysis, up to 100 weeks
  Disease signal detection quantification within each disease cohort, compared to normal controls.
Test performance measures | From date of enrollment to the end of sample analysis, up to 100 weeks
  Sensitivity and specificity/false-positive rate

CONTACTS AND LOCATIONS:
Overall Officials: John Spinosa, MD, PhD, Principal Investigator — Luventix, Inc.
Locations (4):
- United States (4):
  - Unio Health Partners (Gastroenterology), Encinitas, California
  - Digestive Health Associates, Santa Monica, California
  - Westside Gastro Care, Santa Monica, California
  - Bass Medical Group (Gastroenterology), Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasikanti KK, Ho PC, Chan EC. Gas chromatography/mass spectrometry in metabolic profiling of biological fluids. J Chromatogr B Analyt Technol Biomed Life Sci. 2008 Aug 15;871(2):202-11. doi: 10.1016/j.jchromb.2008.04.033. Epub 2008 Apr 29. PMID 18479983
- [Background] Dinges SS, Hohm A, Vandergrift LA, Nowak J, Habbel P, Kaltashov IA, Cheng LL. Cancer metabolomic markers in urine: evidence, techniques and recommendations. Nat Rev Urol. 2019 Jun;16(6):339-362. doi: 10.1038/s41585-019-0185-3. PMID 31092915
- [Background] Wittmann BM, Stirdivant SM, Mitchell MW, Wulff JE, McDunn JE, Li Z, Dennis-Barrie A, Neri BP, Milburn MV, Lotan Y, Wolfert RL. Bladder cancer biomarker discovery using global metabolomic profiling of urine. PLoS One. 2014 Dec 26;9(12):e115870. doi: 10.1371/journal.pone.0115870. eCollection 2014. PMID 25541698
- [Background] Fan J, Hong J, Hu JD, Chen JL. Ion chromatography based urine amino Acid profiling applied for diagnosis of gastric cancer. Gastroenterol Res Pract. 2012;2012:474907. doi: 10.1155/2012/474907. Epub 2012 Jul 25. PMID 22888338
- [Background] Issaq HJ, Nativ O, Waybright T, Luke B, Veenstra TD, Issaq EJ, Kravstov A, Mullerad M. Detection of bladder cancer in human urine by metabolomic profiling using high performance liquid chromatography/mass spectrometry. J Urol. 2008 Jun;179(6):2422-6. doi: 10.1016/j.juro.2008.01.084. Epub 2008 Apr 23. PMID 18433783
- See also: Related Info — https://www.luventix.com